CLINICAL TRIAL: NCT02328560
Title: Impact of the Paramedic Announced Consultation on the Use of Patient Care With Cancer and Treated With Chemotherapy
Acronym: ANNONCEP
Status: Terminated | Type: Observational
Why Stopped: Loss of recrutement
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: ANNONCEP
Record Dates: First submitted 2014-12-10; First posted 2014-12-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-02

CONDITIONS: Solid or Lymphoid Malignant Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Paramedical ad consultation: Monitoring will be the same in the 2 groups; That paramedical consultation announcement is made in current practice.
- No paramedical ad consultation: Monitoring will be the same in the 2 groups

SUMMARY:
The project aims primarily to measure the expected paramedic consultation announcement benefits for the patient, at different levels. It will measure improvements in the management of patients treated with chemotherapy. Indeed, paramedical consultation ad aims to provide a better understanding of the disease and treatment incurred, which should lead to the implementation of joint strategies between the healthcare team and the patient to prevent the effects of and treatment of the disease by the patient and caregivers.

This improvement is to promote the fair treatment by reducing patient anxiety and / or carers and involving them in the management of their disease. In this context, it is shown a profit of paramedical consultation for the patient, it will work, based on the recommendations of the Cancer Plan, strengthen the need to routinely offer paramedic Ad consultation.

This work should also help measure the impact of ad paramedical consultation on optimizing care consumption off-line therapy and to assess the associated costs.

For patients who received paramedic ad or not consultation, it will therefore be of particular compare intercurrent hospitalizations, commuting structure of care, the number of consultations with the doctor, the reports of cure, additional biological monitoring or other health care consumption.

With the participation of several centers in the fight against cancer, this study will provide valuable information on the practice of paramedical consultation ad in several tumor sites.

It will objectify the benefit provided by the Medical device announcement for both patients and the organization and use of care prerequisite to encourage better integration of this device in the course of patient care, the consultation paramedical ad remaining poorly understood by many health professionals.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age <75 years;
* WHO ≤ 1;
* Patients with cancer and candidate for chemotherapy treatment of first intention;
* Solid or lymphoid malignant disease pathology for which chemotherapy is given intravenously;
* Patient affiliated to a social security scheme;
* Mastery of the French language;
* Informed Consent and signed;
* In the first cohort, patients will have received paramedical consultation announcement in the days preceding the first cycle of chemotherapy;
* In the second cohort, patients have not received paramedical consultation announcement.

Exclusion Criteria:

* Patient deprived of liberty, under guardianship;
* Any medical or psychological condition associated that could compromise the patient's ability to participate in the study;
* Exclusive Oral Chemotherapy;
* Exclusive Targeted therapy;
* Targeted therapy to be introduced during chemotherapy;
* Presence of cerebral localization;
* Pain requiring analgesics bearing 3;
* Patient in medical and social structure;
* Inability to submit to medical monitoring test for geographical, social or psychological reasons;
* Rare Cancers making matching difficult (sarcomas of soft tissue and internal organs, malignant neuroendocrine tumors sporadic and hereditary rare ...)
* Inclusion in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment with first-line IV chemotherapy
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Care consumption | Up to 18 weeks
  Compare among patients candidates for chemotherapy treatment IV first line, the proportions of patients who need more care than anticipated during the first cycle of chemotherapy among patients who have had paramedical announcement of consultation and those who have not had.

SECONDARY OUTCOMES:
Hospital costs | Up to 18 weeks
  Evaluate and compare between the 2 groups the total hospital costs
Number of patients with adverse events | Up to 18 weeks
  Evaluate and compare between the 2 groups the health care consumption and side effects of chemotherapy
Satisfaction measured by self-administered questionnaires | Up to 18 weeks
  Evaluate and compare between the 2 groups patient and physicians satisfaction
Anxiety and depression measured by HADS scale | Inclusion
  Compare baseline characteristics of the 2 groups (anxiety and depression)

CONTACTS AND LOCATIONS:
Overall Officials: François GERNIER, health executive, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François BACLESSE, Caen, France